CLINICAL TRIAL: NCT01418664
Title: Prevention of Adverse Pregnancy Outcome With Vitamin D Supplementation During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Nazli Hossain, associate professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 786; other Grant (Other Grant/Funding Number: Pakistan Medical Research Council)
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Pregnancy
Keywords: vitamin D; adverse pregnancy outcome; Pakistan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Active Comparator): Each woman in above group will recieve in addition to routine ferrous sulphate and calcium lactate, 4000IU of vitamin D
  Interventions: Dietary Supplement: D Max drops
- control group (No Intervention): Women in this group will recieve ferrous sulphate and calcium lactate

INTERVENTIONS:
Dietary Supplement: D Max drops — Women in study arm will be cases, and will recieve ferrous sulphate and calcium lactate, along with 4000IU D Max drops
  Arms: Study group

SUMMARY:
We hypothesized that vitamin D supplementation during pregnancy can prevent adverse pregnancy outcome.

DETAILED DESCRIPTION:
Vitamin D deficiency has been associated with many chronic diseases. These include cardiovascular diseases, diabetes mellitus, multiple sclerosis, breast and prostate cancers. Recently, its role in pregnancy has been explored. Vitamin D deficiency has been found to be associated with adverse pregnancy outcome. These include pre eclampsia, gestational diabetes mellitus, preterm labor and low birth weight.

Bodnar et al, evaluated role of vitamin D deficiency during pregnancy in PE in a nested case control study. The investigators looked at the role of vitamin D at gestational age of < 22 weeks. Women who developed PE were found to have low levels of vitamin D. These women had serum levels of vitamin D < 15 ng/ml, were supplemented during pregnancy with prenatal vitamins, were still found to have 5 fold greater chances of developing PE (adjusted odds ratio, 5.0; 95% confidence interval, 1.7-14.1).Children of above group of women were also found to have low levels of vitamin D. The authors concluded that vitamin D deficiency may be an independent factor for the development of PE.(1)

In an epidemiological study from Norway, involving 23,423 primigravidae, the rsik of PE was found to be 27% greater in women who did not receive D supplements, compared to women who received 10-15µg/day of vitamin D(2).

Circulating levels of 1-25(OH) have been found to be low in women with PE.(3) This has been attributed to reduced expression and activity of 1α-hydroxylase in human placenta from preeclamptic pregnancies.(4) This association with PE has also been found to be influenced by VEGF (Vascular endothelial growth factor). Active forms of vitamin D have been found to increase the expression of VEGF , and its release in vascular smooth cells, in in-vitro studies.(5)

Vitamin D deficiency has also been associated with small for gestational age (SGA) (6) The difference has been found to be more subtle for Caucasians as compared to African-Americans in West. The investigators showed a U shaped association between D levels and SGA. After confounder adjustment, compared with serum 25(OH)D 37.5-75 nmol/L, SGA odds ratios (95% CI) for levels <37.5 and >75 nmol/L were 7.5 (1.8, 31.9) and 2.1 (1.2, 3.8), respectively. In a similar study by Brooke, among Asian women resident in UK, vitamin D supplementation with 1000IU in third trimester, compared with placebo, was associated with decreased incidence of small for gestational age (15% versus 29%). Investigators suggested supplementation with vitamin D among Asians living in UK.(7)

Vitamin D deficiency has been related to gestational diabetes mellitus (GDM) in pregnant women. Zhang et al, found that vitamin D deficiency in early pregnancy is linked with increased risk for GDM. Vitamin D deficiency was associated with a 2.66-fold (OR (95% CI): 2.66 (1.01-7.02)) increased GDM risk. Moreover, each 5 ng/ml decrease in 25-[OH] D concentrations was related to a 1.29-fold increase in GDM risk (OR (95% CI): 1.29 (1.05-1.60)).(8) Similarly, in an Iranian study, women who were found to have GDM, were found to have lower levels of serum 1,25 (OH), as compared to normoglycemic women. (9) Serum levels of <12 nmol/L were found associated with GDM. This may be linked to the fact that 1,25(OH) stimulates insulin secretion.

Vitamin D deficiency has also been linked to increased risk for cesarean section. In a study of 253 women, who underwent cesarean section, multivariable logistic regression analysis controlling for race, age, education level, insurance status, and alcohol use, women with 25(OH)D less than 37.5 nmol/liter were almost 4 times as likely to have a cesarean than women with 25(OH)D 37.5 nmol/liter or greater (adjusted odds ratio 3.84; 95% confidence interval 1.71 to 8.62).(10) Poor muscular performance due to vitamin D deficiency may be the reason for the increased cesarean section rate.

Preterm labor, is the other adverse pregnancy outcome, which is thought to be affected by maternal serum levels of 1,25(OH). In a recently concluded RCT, a comparison was made between 400IU, 2000IU and 4000IU of daily supplementation with vitamin D. Women who were prescribed highest doses had significant less chances of spontaneous preterm birth at < 37 and at < 32 weeks.(11) Inflammation plays a key role in the etiology of preterm labor. And vitamin D is known to influence the production of inflammatory mediators like interleukin 1, interleukin -6 and tumor necrosis factor by macrophages.(12) This may be a reason for decreased incidence of preterm birth in women who received vitamin D supplementation.

Birth weight of newborn is also affected by maternal serum D levels. In a study from neighboring Iran, of 449 women, birth weight, length and apgar score were significantly better in women who took diet adequate in calcium and vitamin D.(13) Vitamin D supplementation during pregnancy leads to increased calcium stores in infants and improved weight gain as well. Levels < 25ng/ml are associated with rickets and osteomalacia. There is positive correlation between maternal and neonatal cord levels of vitamin D. This relationship has also been shown in studies from other part of world. (14-16)This indicates that these newborns are entering the world, with deficiency of vitamin D, which starts in utero. Apart from affecting skeletal development, it also affects the innate immune system of newborn. In a case-control study, children who were deficient in vitamin D were found to be more prone to acute respiratory tract infections. The mean serum 25(OH)D concentrations in the study group newborns were lower than those of the control group (9.12+/-8.88 ng/ml and 16.33+/-13.42 ng/ml, respectively) (P=0.011). (17) It has been observed that infants born to D replete mothers will become D deficient, 8 weeks after birth, unless they are supplemented with vitamin D. In an earlier cross sectional study, from Karachi city Atiq M, had found low levels of vitamin D in newborns who were breastfed. The age group was from 6 weeks to 11 months. Thirty-four (48%) mothers and 37 (52%) infants had levels less than 25 nmol/ L (i.e. <10ng/ml). The investigators found a significant correlation between serum 25(OH)D levels of infants under three months of age and their mothers (p<0.01).(18) Though this study was carried out in a private university hospital, where majority of mothers belonged to upper socio economic class.

Content of vitamin D in breast milk is dependant upon the serum levels in mothers. Supplementation of lactating mothers has been recommended to avoid deficiency in newborn, but is not a norm in our practice. There is also increased motivation for exclusive breast feeding for the first 4-6 months in our society. Hence with prevalence of vitamin D deficiency as high as 90% in our population (data submitted for publication), our newborns are more at risk for vitamin D deficient rickets

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending antenatal clinic at ≤ 20 weeks of gestation
* Normoglycemic, normotensive at the time of antenatal booking

Exclusion Criteria:

* Multiple pregnancy
* H/O hypertensive disorders in previous pregnancy
* Known diabetic or h/o gestational diabetes in previous pregnancy
* H/O endocrine disorders ( thyroid, parathyroid dysfunction)
* Chronic renal diseases
* Tuberculosis
* Breast feeding (current)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2010-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Prevention of adverse pregnancy outcome, viz preeclampsia, small for gestational age (SGA), preterm labor | 18 months

SECONDARY OUTCOMES:
Cord levels and maternal serum levels of 1,25(OH), after supplementation at the time of delivery. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Nazli Hossain, MBBS, FCPS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data has been published

REFERENCES:
- [Derived] Finkelstein JL, Cuthbert A, Weeks J, Venkatramanan S, Larvie DY, De-Regil LM, Garcia-Casal MN. Daily oral iron supplementation during pregnancy. Cochrane Database Syst Rev. 2024 Aug 15;8(8):CD004736. doi: 10.1002/14651858.CD004736.pub6. PMID 39145520
- [Derived] Hossain N, Kanani FH, Ramzan S, Kausar R, Ayaz S, Khanani R, Pal L. Obstetric and neonatal outcomes of maternal vitamin D supplementation: results of an open-label, randomized controlled trial of antenatal vitamin D supplementation in Pakistani women. J Clin Endocrinol Metab. 2014 Jul;99(7):2448-55. doi: 10.1210/jc.2013-3491. Epub 2014 Mar 19. PMID 24646102